CLINICAL TRIAL: NCT06535399
Title: A Phase 1, Multi-center, Open-label, Single-dose Study to Assess the Pharmacokinetics and Safety of Golcadomide (BMS-986369) in Healthy Participants and Participants With Moderate and Severe Hepatic Impairment
Brief Title: Study to Assess Drug Levels and Safety of Golcadomide (BMS-986369) in Healthy Participants and Participants With Different Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA073-1028
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Healthy Volunteers; Pharmacokinetics; Liver Diseases; Moderate and Severe Hepatic Impairment; BMS-986369; CC-99282; Hepatic Impairment; Golcadomide
MeSH Terms: conditions — Liver Diseases; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: BMS-986369 Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: BMS-986369
- Group B: BMS-986369 Severe Hepatic Impairment (Experimental)
  Interventions: Drug: BMS-986369
- Group C: BMS-986369 Normal Hepatic Function (Experimental)
  Interventions: Drug: BMS-986369

INTERVENTIONS:
Drug: BMS-986369 — Specified dose on specified days
  Other Names: Golcadomide

SUMMARY:
The purpose of this study is to assess the drug levels and safety of golcadomide (BMS-986369) in adult participants with moderate and severe Hepatic Impairment (HI), and in matched healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria for all Participants (Group A, Group B, Group C):

* Body mass index (BMI) between 18 and 40 kg/m^2 (inclusive), and body weight ≥ 50 kg.

Inclusion Criteria for Participants with Moderate or Severe Hepatic Impairment (Group A and Group B):

* Participants have moderate HI (Group A), severe HI (Group B) or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
* Participants have moderate (Group A) or severe (Group B) HI as defined by National Cancer Institute-Organ Dysfunction Working Group (NCI-ODWG) criteria.

Inclusion Criteria for a Matched Healthy Participant (Group C):

* Participants must have liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions as agreed by the investigator and the Sponsor Medical Monitor.
* Participants must be free of any clinically significant disease that would interfere with the study evaluations.

Exclusion Criteria for all Participants (Group A, Group B, and Group C):

* Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism, and excretion (ADME).
* History of major surgery within 8 weeks before the study intervention administration.
* Any other clinically significant medical, psychiatric, and/or social reason, or other active issues, as determined by the investigator.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 44 days
Time of maximum observed plasma concentration (Tmax) | Up to approximately 44 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to approximately 44 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 44 days
Incidence of serious adverse events (SAEs) | Up to approximately 44 days
Number of participants with physical examination abnormalities | Up to approximately 44 days
Number of participants with vital sign abnormalities | Up to approximately 44 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to approximately 44 days
Number of participants with clinical safety laboratory test abnormalities | Up to approximately 44 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 0001, Chandler, Arizona
  - Local Institution - 0002, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com